CLINICAL TRIAL: NCT03760328
Title: Effect of Upper Airway Stimulation: A Randomized Controlled Crossover Study
Brief Title: Effect of Upper Airway Stimulation in Patients With Obstructive Sleep Apnea
Acronym: EFFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Universitätsmedizin Mannheim (Other); University of Luebeck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EFFECT
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multi-center, randomized, crossover study, conducted under a common protocol. Subjects will be enrolled after they have been implanted and using the Inspire therapy (Inspire II/IV, Inspire Medical Systems, Maple Grove, USA) for at least six months. Participants will be randomized to one of two groups: therapeutic stimulation or sham stimulation. During the second phase of the study therapy settings of the stimulation system will be adjusted to crossover.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the subject nor the investigator or Outcomes Assessor (double-blinded) will know the outcome of the randomization until after the subject has fulfilled and completed all study requirements at the end of the visit 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic stimulation (Active Comparator): Therapeutic Stimulation: optimal therapy setting for home use
  Interventions: Device: Upper Airway Stimulation
- sham stimulation (Sham Comparator): Sham Stimulation (Control Group): stimulation voltage programmed at 0.1 volts
  Interventions: Device: Upper Airway Stimulation

INTERVENTIONS:
Device: Upper Airway Stimulation — hypoglossal nerve stimulation by using a breathing cycle depended stimulation system of the upper airway
  Other Names: Inspire

SUMMARY:
Upper Airway Stimulation is a new therapy, which is available for patients with obstructive sleep apnea, who are non-compliant to the standard treatment continuous positive airway pressure (CPAP) therapy. This study is a prospective, multi-center, double-blinded, randomized crossover study conducted under a common protocol. The study visits include baseline with an in-laboratory polysomnography (PSG) after six months of therapy usage, followed by visits and in-lab PSGs at 1 and 2-weeks where the Therapy stimulation will be changed at each, according to randomization. The objective of this randomized controlled crossover study is to assess treatment effect of Inspire UAS in patients at different time points with two different therapy settings. This study will provide additional clinical evidence of Inspire UAS for treatment of moderate to severe OSA using a randomized controlled crossover trial design.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is characterized by recurrent episodes of airflow obstruction in the upper airway that results in oxygen desaturations and arousal from sleep. The most common symptom of OSA is excessive daytime sleepiness. Recent studies have also shown clear association of OSA with the development of obesity, hypertension diabetes mellitus, and congestive heart failure. Approximately 13% men and 6% women have moderate to severe OSA (apnea hypopnea index, AHI ≥ 15) in the US.

The efficacy of therapies for OSA, and in particular, continuous positive airway pressure (CPAP) has been limited due to patient intolerance, poor patient selection, or limited response to the therapy.

The Inspire Upper Airway Stimulation (UAS) system is intended to prevent upper airway obstruction by stimulating the hypoglossal nerve synchronous with respiration [7].

The Inspire system is comprised of the following components:

* Inspire Upper Airway Stimulator (Implantable Pulse Generator (IPG))
* Inspire Stimulation Lead
* Inspire Sensing Lead
* External programmers used with the system are:

  * Inspire Programmer (physician programmer)
  * Inspire Patient Programmer (patient remote)

The Inspire system received CE Mark in 2010 (CE Certificate No. 562872) providing the regulatory authority to provide the device in a commercial setting. Furthermore, this study will be conducted within the CE marked intended use of the Inspire system and will not involve any additional stressful or invasive tests.

The objective of this randomized controlled crossover study is to assess treatment effect of Inspire UAS in patients at different time points with two different therapy settings. This study will provide additional clinical evidence of Inspire UAS for treatment of moderate to severe OSA using a randomized controlled crossover trial design.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy subjects that are at least 18 years old and:

  1. Have been implanted and using the Inspire Therapy for at least six months
  2. Willing and capable to undergo three in-lab PSGs in a one-month timeframe
  3. Willing and capable of having reduced Inspire stimulation for one week
  4. Willing and capable of providing informed consent

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this clinical investigation:

  1. Unwilling to complete three in-lab PSGs within a 1-month timeframe
  2. Any other reason the investigator deems subject is unfit for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in AHI from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  Apnea Hypopnea Index (AHI) is a measure of OSA severity. The AHI in this study will be determined by the AHI score at Visit 1 and Visit 2 compared with the baseline score.
Change in ESS from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  The Epworth Sleepiness Scale (ESS) is a validated instruction that rates a subject's daytime sleepiness. The ESS efficacy endpoint will be determined by the ESS score at Visit 1 and Visit 2 as compared to baseline.

SECONDARY OUTCOMES:
Change in FOSQ from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  The Functional Outcomes of Sleep Questionnaire (FOSQ) is a validated instrument to assess the effect of a subject's daytime sleepiness on activities of ordinary living. The FOSQ endpoint will be determined by the FOSQ score at Visit 1 and Visit 2 as compared to baseline.
Change in Snoring Intensity from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  Snoring Intensity will be measured by using a visual analoge scale from 0 (no snoring) to 10 (heavy snoring). The snoring intensity endpoint will be determined by the visual analogue scale at Visit 1 and Visit 2 as compared to baseline.
Therapy Adherence | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  Therapy use, reported as hours of use per week, is record by Inspire device and can be collected upon interrogation of the device in the clinic. This value can be used to quantify device use and adherence over the investigated time period.
Change in ODI from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  Oxygen Desaturation Index (ODI) is a measure of OSA severity. The ODI will be determined by the ODI score at Visit 1 and Visit 2 as compared with to baseline
Change in Clinical Global Impression (CGI-I) from Baseline to Visit 1 and Visit 2 | Baseline through Visit 1 (1 week) and Visit 2 (2 weeks)
  The CGI-I is a seven point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Heiser, M.D., Principal Investigator — Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Department of Ear Nose Throat, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steffen A, Moritz FJ, Konig IR, Suurna MV, Bruggemann N. Electric field aspects in hypoglossal nerve stimulation for obstructive sleep apnea: A bilateral electrophysiological evaluation of unilateral electrode configuration changes. J Sleep Res. 2023 Feb;32(1):e13592. doi: 10.1111/jsr.13592. Epub 2022 May 21. PMID 35596592
- See also: Homepage for Department — http://www.schlaf-hno.de